CLINICAL TRIAL: NCT00893321
Title: Comparison of Inferior Oblique Muscle Recession and Myectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8701
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Inferior Oblique Muscle Overactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inferior Oblique Muscle Recession and Myectomy (Other)
  Interventions: Procedure: Inferior Oblique Muscle Recession and Myectomy

INTERVENTIONS:
Procedure: Inferior Oblique Muscle Recession and Myectomy

SUMMARY:
The purpose of this study is to compare muscle recession and myectomy on inferior oblique muscle overactivity.

ELIGIBILITY:
Inclusion Criteria:

* Overactivity of Inferior Oblique Muscle >= 2

Exclusion Criteria:

* Nystagmus
* History of vertical muscle operation
* Mechanical limitation
* Eye disease
* Paralysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-05 (Estimated); Study Completion 2009-09 (Estimated)